CLINICAL TRIAL: NCT02754167
Title: Phase Ib Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of the Hepcidin Antagonist PRS-080#022-DP in Anemic Chronic Kidney Disease Patients Undergoing Hemodialysis
Brief Title: Phase Ib Study to Evaluate PRS-080 in Anemic Chronic Kidney Disease Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pieris Pharmaceuticals GmbH (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCS_02_15
Record Dates: First submitted 2016-04-14; First posted 2016-04-28 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Anemia of Chronic Kidney Disease
Keywords: Hepcidin; hemoglobin; iron; anemia of chronic disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRS-080#022-DP (Experimental): Hepcidin antagonist, single administration, ascending doses
  Interventions: Biological: PRS-080#022-DP
- PRS-080-Placebo#001 (Placebo Comparator): Comparator treatment, single administration
  Interventions: Biological: PRS-080-Placebo#001

INTERVENTIONS:
Biological: PRS-080#022-DP — Hepcidin antagonism to mobilize iron and to treat anemia
  Other Names: PRS-080
  Arms: PRS-080#022-DP
Biological: PRS-080-Placebo#001 — Placebo comparator
  Other Names: Placebo
  Arms: PRS-080-Placebo#001

SUMMARY:
Anticalins® are engineered human proteins that are able to bind specific target molecules. The Anticalin PRS-080#022-DP to be investigated in this study is directed against hepcidin and is intended for the treatment of anemia of chronic disease. This Phase Ib study shall investigate the safety, pharmacokinetics and pharmacodynamics of a single administration of PRS-080#022-DP in anemic stage 5 chronic kidney disease patients undergoing hemodialysis.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled, single ascending dose phase Ib study in anemic stage 5 chronic kidney disease patients requiring hemodialysis. Eligible subjects will undergo screening assessments and PRS-080#22-DP will be administered by intravenous infusion. The study will consist of 3 dose cohorts of 2 mg/kg, 4 mg/kg, and 8 mg/kg body weight with 8 subjects in each cohort. Using a standard 6+2 design, 6 subjects in each cohort will be randomized to PRS-080#022-DP and 2 subjects in each cohort will be randomized to placebo. The decision to escalate the dose will be based on an interim analysis of clinical safety and safety laboratory data. Safety and tolerability, pharmacokinetics, pharmacodynamics as well as potential immunogenicity will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage 5 chronic kidney disease having been on hemodialysis for at least 90 days
* Patients being on stable erythropoiesis-stimulating agent (ESA) dose
* Hemoglobin (Hb) 9 - 11 g/dL
* Ferritin ≥ 300 ng/mL.
* Transferrin saturation (TSAT) ≤ 30%
* Hepcidin 5 - 50 nmol/L

Exclusion Criteria:

* Anemia due to causes other than chronic kidney disease, including hemoglobinopathies, hemolytic anemias, myelodysplasia or malignancy
* Blood transfusion within 2 months before administration of study medication.
* Iron treatment from 1 week before study medication administration until 1 week after study medication administration.
* Previous enrollment in this study
* Current or previous (within 60 days before study medication administration) treatment with another investigational drug and/or medical device or participation in another clinical study.
* Pregnancy or breast-feeding women of child bearing age.
* Known allergy to any component of the PRS-080#022-DP formulation
* Positive for hepatitis B surface antigen, anti-hepatitis C virus antibody, or human immunodeficiency virus
* Planned surgery during the study period
* Unwilling or unable to comply with the protocol, in the judgment of the investigator
* Unstable angina, myocardial infarction, percutaneous transluminal coronary angioplasty/stents, apoplexy or coronary artery bypass grafting <3 months prior screening.
* Congestive heart failure: New York Heart Association Class III or IV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events | 28 days
  Composite measure including signs and symptoms, changes from baseline heart rate and blood pressure, ECG, body temperature, respiratory rate clinical chemistry and hematology

SECONDARY OUTCOMES:
Pharmacokinetics of PRS-080#022 | 28 days
  Area under the plasma concentration versus time curve (AUC) of PRS-080 in plasma
Effects of PRS-080#022 on serum iron | 28 days
  Changes in total serum iron concentration compared to baseline
Effects of PRS-080#022 on ferritin | 28 days
  Changes in serum ferritin concentration compared to baseline
Effects of PRS-080#022 on transferrin saturation | 28 days
  Changes in serum transferrin saturation compared to baseline
Effect of PRS-080#022 on hepcidin concentrations in plasma | 28 days
  Changes in hepcidin concentration compared to baseline
Number of patients developing anti-drug antibodies | 28 days
  Number of patients with antibodies against PRS-080#022 at day 28 compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Lutz Renders, Prof. MD, Principal Investigator — Technical University, Munich
Locations (2):
- Germany (2):
  - St. Joseph Krankenhaus, Berlin
  - Technical University, Medical Department, Munich

IPD SHARING:
Plan to Share IPD: No